CLINICAL TRIAL: NCT03404544
Title: Evaluation of the Impact of Carbetocin Administration (Bolus Versus Infusion) on Heart Rate and Other Hemodynamic Parameters.
Brief Title: Impact of Carbetocin Administration on Heart Rate When Given as an Infusion Versus as a Bolus.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Philippe Richebe, Professor of Anesthesiology and Pain Medicine, Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2018-1213
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Cesarean Section Complications; Hemodynamic Instability

STUDY DESIGN:
Intervention Model Description: Prevention of hemodynamic carbetocin-induced side effects when the study drug carbetocin 100 mcg intravenous is given as an infusion over 10 minutes versus a single shot rapid bolus (same dose). Two syringes per subject will be prepared by the research nurse :
  1. one 3 ml syringe containing 1 ml of either carbetocin 100 mcg or normal saline (according to the patient's study group);
  2. one 10 ml syringe containing carbetocin 100 mcg (1 ml) diluted with 9 ml of normal saline for a total volume of 10 ml, or 10 ml of normal saline (according to the patient's study group).
  The volume in the 3 ml syringe will be injected as an IV push bolus after cord clamping and the volume in the 10 ml syringe will be infused over 10 minutes at cord clamping. The study subject, the attending anesthesiologist and the anesthesiologist collecting intraoperative data will be blinded to patient group allocation. The research nurse will not be blinded to patient group allocation.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Only the clinical nurse won't be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbetocin bolus (Active Comparator): Patients in this arm will receive both syringes : the 3 ml and the 10 ml. The carbetocin 100 mcg will be in the 3 ml syringe over 2 sec and the 10 ml syringe will contain only normal saline given as infusion over 10 min.
  Interventions: Drug: Carbetocin bolus
- Carbetocin infusion (Experimental): Patients in this arm will receive both syringes : the 3 ml and the 10 ml. The carbetocin 100 mcg will be in the 10 ml syringe as an infusion over 10min and the 3 ml syringe will contain only normal saline given iv over 2 sec as a bolus.
  Interventions: Drug: Carbetocin infusion

INTERVENTIONS:
Drug: Carbetocin bolus — Carbetocin 100 mcg intravenous as a bolus (less than 2 sec)
  Other Names: Duratocin
  Arms: Carbetocin bolus
Drug: Carbetocin infusion — Carbetocin 100 mcg intravenous as a 10 minutes infusion
  Other Names: Duratocin
  Arms: Carbetocin infusion

SUMMARY:
Prospective, randomized and controlled study who will be conducted at Maisonneuve-Rosemont hospital with the following objectives:

To determine if an infusion of carbetocin over 10 minutes will reduce hemodynamic side effects, especially the peak of heart rate, in comparison to a rapid intravenous bolus (less than 2 seconds).

To determine if an infusion of carbetocin will reduce the other side effects of duratocin in comparison to a rapid intravenous bolus.

Study plans to enroll 70 adult patients scheduled to undergo elective cesarean delivery under spinal anesthesia.

Half of the patient will receive Carbetocin 100 mcg intravenous as a bolus (less than 2 seconds) and the other half will receive Carbetocin 100 mcg intravenous infusion over 10 minutes.

DETAILED DESCRIPTION:
The purpose of this prospective pragmatic study is to determine if an infusion of carbetocin over 10 minutes will reduce hemodynamic compromise in comparison to a rapid intravenous bolus (less than 2 seconds) during elective cesarean delivery under spinal anesthesia.

In this prospective, randomized and controlled study, each parturient will enter the operating room on the day scheduled for there surgery. All the classic monitors will be installed, along with the Edwards (Clear sight system).

Each patient will receive an antacid prophylaxis of 30 ml of sodium citrate per mouth 30 min before surgery. Baseline measures of BP (blood pressure), HR (Heart Rate), O2 Arterial Saturation will be taken before entering in the operating room, in a calm environment.

The anesthetic technique will be standardized. Spinal anesthesia will be performed in the sitting position by the anesthesiologist in charge of the patient, with the local anesthetic injected between L2 to L5 spinal level. The anesthetic solution will consist of hyperbaric bupivacaine 0.75% 10.5 mg, fentanyl 15 μg, and morphine 150 μg with a Whitacre needle 25G ou 27G. Then, the patient will be immediately placed in the supine position, with a cushion under their right hip or a left lateral tilt. Antibiotic prophylaxis will be administered to each patient before incision.

Each patient included in the study will have a phenylephrine infusion of 0.5 mcg/kg/min (lean body weight) started immediately after the injection of local anesthetic. A bolus of phenylephrine 1.5 mcg/kg (lean body weight) will be administered in case of a hypotensive episode. A hypotensive episode will be defined as 2 consecutive Systolic BP (SBP) measurements less than 20% below the baseline value. The treatment of hypotension consists of Phenylephrine 1.5 mcg/kg intravenous bolus will be administered if HR > 55 bpm or Ephedrine 5 mg intravenous bolus if HR is < 55 bpm. If only the HR is < 55 bpm, but SBP is normal, Glycopyrrolate 0.2 mg intravenous bolus will be administered and the patient will be excluded. In the case of a hypertensive episode, where systolic BP is > 120% Baseline value, treatment will consist of a decrease in the phenylephrine infusion rate by 0.2 mcg/kg/min.

In addition, each patient included in the study will receive an intravenous volume co-load of 1000 ml of Lactate Ringer administered under pressure in 5 to 10 minutes immediately after installing the intravenous catheter, and before and during the spinal anesthesia. Then, an infusion of Lactate Ringer at 300 mL/h will begin.

Surgery will begin after the confirmation of a sensory block to cold stimulus at the T4 level.

Data collection will be realized with the Edwards monitor, and HR (Heart Rate), BP (Blood Pressure), SV (Stroke Volume), SVV (Stroke Volume Variation), CO (Cardiac Output), SVR will be taken continuously every 20 seconds. HR, BP, and pulse oxymetry values will also be measured every 2.5 minutes with the applied standard monitoring, from the intrathecal injection of the local anesthetic until the neonate is born. After the injection of the study drug, those values will be measured every minute for 20 minutes (All these data are electronically recorded every 5 seconds). Hemodynamic values recorded at skin incision will be used as baseline values for comparison with hemodynamic measurements recorded over the 20 minutes following the beginning of study drug infusion.

All subjects will receive Metoclopramide 10mg intravenously at the induction of anesthesia for anti-emesis prophylaxis and Ondansetron 4 mg IV for intraoperative treatment of nausea and/or vomiting.

Prevention of post-partum hemorrhage will be with the study drug carbetocin 100 mcg given intravenously, either as a bolus or an infusion over 10 min, depending on the randomization. Two syringes per subject will be prepared by the research nurse :

1. one 3 ml syringe containing 1 ml of either carbetocin 100 mcg or normal saline same volume (according to the patient's study group);
2. one 10 ml syringe containing carbetocin 100 mcg (1 ml) diluted with 9 ml of normal saline for a total volume of 10 ml, or 10 ml of normal saline (according to the patient's study group).

The volume in the 3 ml syringe will be injected as an IV push bolus after cord clamping and the volume in the 10 ml syringe will be infused over 10 minutes at cord clamping. The study subject, the attending anesthesiologist and the anesthesiologist collecting intraoperative data will be blinded to patient group allocation. The research nurse will not be blinded to patient group allocation.

The uterine repair will be done in situ and not by exteriorization. In the eventuality that the attending obstetrician proceeded to exteriorization of the uterus for safety reasons, the patient would then be excluded from the study.

Uterine tone will be assessed by the attending obstetrician as adequate or inadequate at the end of the 10 minutes study drug infusion. If uterine tone is judged inadequate, patient care will be carried on by the attending anesthesiologist and obstetrician according to best clinical practice guidelines. These patients will be excluded from the study.

The data collection will be achieved by the ClearSight (Edwards) system. It will start before the uterine incision and will continue until 20 minutes after the beginning of the carbetocin (or normal saline) 10 minutes infusion.

ELIGIBILITY:
Inclusion Criteria:

* Elective caesarean delivery
* 37 weeks or more of gestation
* ASA status I or II
* Patients > 18 years old
* Spinal anesthesia

Non-Inclusion Criteria:

* Multiple gestation
* Morbid obesity (BMI > 40 at first prenatal medical visit)
* Coagulopathy
* Active labour
* Polyhydramnios
* Leiomyoma/Uterine fibroma
* Hypotensive illness/Pre-eclampsia/Eclampsia
* Placenta accreta/Previa
* Cardiopathy of any kind
* Patient on medication affecting hemodynamics (ex. B-blocker, CCG, antihypertensive, etc)
* Emergent cesarean delivery
* Contra-indications to spinal anesthesia
* General anesthesia for cesarean delivery
* Known allergy to carbetocin
* Patient refusal

Exclusion criteria

* Patient who receives iv ephedrine or glycopyrrolate during the study period
* Administration of a second dose of carbetocin or other uterotonic agent.
* Onset of post-partum hemorrhage defined as blood loss > 1000 ml or uncontrolled bleeding after delivery of the baby.
* Patient who needs an exteriorization of the uterus for repair following caesarean delivery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Delta Heart Rate | From the administration of the drug study every 20 secondes until 20 minutes after the drug injection for each patient.
  To compare the variation of HR (delta heart rate) after the administration of Carbetocin when administered in Infusion vs Bolus, in patients with elective Caesarian under regional anesthesia.

SECONDARY OUTCOMES:
Delta Stroke Volume | From the administration of the drug study every 20 secondes until 20 minutes after the drug injection for each patient.
  To compare the variation of Stroke Volume (delta stroke volume) after the administration of Carbetocin when administered in Infusion vs Bolus, in patients with elective Caesarian under regional anesthesia.
Delta Stroke Volume Variation | From the administration of the drug study every 20 secondes until 20 minutes after the drug injection for each patient.
  To compare the variation of stroke volume variation in a respiratory cycle (delta stroke volume variation) after the administration of carbetocin in infusion vs bolus in patients with elective Caesarian under regional anesthesia.
Delta Cardiac Output | From the administration of the drug study every 20 secondes until 20 minutes after the drug injection for each patient.
  To compare the variation of cardiac output (delta cardiac output) after the administration of carbetocin in infusion vs bolus in patients with elective Caesarian under regional anesthesia.
Delta Systemic Vascular Resistance | From the administration of the drug study every 20 secondes until 20 minutes after the drug injection for each patient.
  To compare the variation of systemic vascular resistance (delta systemic vascular resistance) after the administration of carbetocin in infusion vs bolus in patients with elective Caesarian under regional anesthesia.
Peak value of Heart Rate | From the administration of the drug study every 20 secondes until 20 minutes after the drug injection for each patient.
  To compare the peak value of Heart Rate after the administration of Carbetocin in the infusion group vs bolus group.
Peak value of Stroke Volume | From the administration of the drug study every 20 secondes until 20 minutes after the drug injection for each patient.
  To compare the peak value of stroke volume after the administration of Carbetocin in the infusion group vs bolus group.
Peak value of Cardiac Output | From the administration of the drug study every 20 secondes until 20 minutes after the drug injection for each patient.
  To compare the peak value of cardiac output after the administration of Carbetocin in the infusion group vs bolus group.
Peak value of Systemic Vascular Resistance | From the administration of the drug study every 20 secondes until 20 minutes after the drug injection for each patient.
  To compare the peak value of Systemic Vascular Resistance after the administration of Carbetocin in the infusion group vs bolus group.
Phenylephrine consomption in the Infusion group VS Bolus group | From the administration of the drug study every 5 minutes until 20 minutes after the drug injection for each patient.
  To compare the phenylephrine consomption after administration of Carbetocin in the Infusion group VS Bolus group.
Area Under the Curve of Heart Rate for Carbetocin Infusion vs Bolus | From the administration of the drug study until 20 minutes after the drug injection for each patient.
  To compare the AUC between the infusion group versus the bolus group for the heart rate
Area Under the Curve of Cardiac Output for Carbetocin Infusion Vs Bolus | From the administration of the drug study until 20 minutes after the drug injection for each patient.
  To compare the AUC between the infusion group versus the bolus group for the Cardiac Output
Area Under the Curve of Phenylephrine consomption for Carbetocin Infusion Vs Bolus | From the administration of the drug study until 20 minutes after the drug injection for each patient.
  To compare the AUC between the infusion group versus the bolus group for the phenylephrine consomption
Amount of time (in minutes) Heart Rate will be at his peak after administration of carbetocin | From the administration of the drug study every 20 secondes until 20 minutes after the drug injection for each patient.
  To compare the amount of time (in minutes) the heart rate will be at his peak after administration of carbetocin in Infusion group Vs Bolus group
Time (bloc of 5 minutes) for the maximal consomption of phenylephrine | From the administration of the drug study every 5 minutes until 20 minutes after the drug injection for each patient.
  To compare the timing (bloc of 5 minutes) for the maximal consomption of phenylephrine after administration of Carbetocin in the Infusion group Vs Bolus group
Incidence of flushing | From the administration of the drug study until 20 minutes after the drug injection for each patient.
  To compare the incidence of flushing (yes or no) after administration of carbetocin in the Infusion group Vs Bolus Group.
Incidence of headache | From the administration of the drug study until 20 minutes after the drug injection for each patient.
  To compare the incidence of flushing (yes or no) after administration of carbetocin in the Infusion group Vs Bolus Group.
Incidence of thoracic pain | From the administration of the drug study until 20 minutes after the drug injection for each patient.
  To compare the incidence of flushing (yes or no) after administration of carbetocin in the Infusion group Vs Bolus Group.
Incidence of abdominal pain | From the administration of the drug study until 20 minutes after the drug injection for each patient.
  To compare the incidence of abdominal pain (yes or no) after administration of carbetocin in the Infusion group Vs Bolus Group.
Incidence of tremulousness | From the administration of the drug study until 20 minutes after the drug injection for each patient.
  To compare the incidence of tremulousness (yes or no) after administration of carbetocin in the Infusion group Vs Bolus Group.
Incidence of dyspnea | From the administration of the drug study until 20 minutes after the drug injection for each patient.
  To compare the incidence of dyspnea (yes or no) after administration of carbetocin in the Infusion group Vs Bolus Group.
Incidence of nausea/vomiting | From the administration of the drug study until 20 minutes after the drug injection for each patient.
  To compare the incidence of nausea/vomiting moderate to severe (scale of PONV) after administration of carbetocin in the Infusion group Vs Bolus Group.

CONTACTS AND LOCATIONS:
Locations (1):
- CIUSSS de l'Est de l'Ile de Montreal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Boisselle ME, Zaphiratos VV, Fortier A, Richebe P, Loubert C. Comparison of carbetocin as a bolus or an infusion with prophylactic phenylephrine on maternal heart rate during Cesarean delivery under spinal anesthesia: a double-blinded randomized controlled trial. Can J Anaesth. 2022 Jun;69(6):715-725. doi: 10.1007/s12630-022-02227-y. Epub 2022 Mar 30. PMID 35352277